CLINICAL TRIAL: NCT06914414
Title: Interventional Neuroradiology Evaluation of a 3D Silicon Flow Model Representing the Aorto Cervicoencephalic Arterial Tree, Enabling the Patient to Simulate the Entire Procedure During the Preoperative Consultation
Brief Title: Impact of Life-size 3D Model on Patient Anxiety During Intracranial Aneurysms Embolization in Interventional Neuroradiology.
Acronym: ANXIFLOW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-0030 chu caen; CHU CAEN (Other: CHU CAEN)
Record Dates: First submitted 2025-03-24; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Aneurysm Unruptured
Keywords: aneurysm; anxiety; flow model
MeSH Terms: conditions — Aneurysm; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): Patient undergoing embolization of an unruptured aneurysm with standard management (medical consultation with the physician) + a paramedical consultation with oral information and explanations by the radiology technician (one week before the procedure)
- Experimental (Experimental): Patient undergoing embolization of unruptured aneurysm with standard management (medical consultation with the physician) + paramedical consultation with oral information and presentation of the flow model by the radiology technician (one week before the procedure)
  Interventions: Procedure: Using the flow model in cerebral aneurysm embolization

INTERVENTIONS:
Procedure: Using the flow model in cerebral aneurysm embolization — Since the 1970s-1980s, surgical techniques for intracranial aneurysms have evolved. In recent years, endovascular embolization of aneurysms has demonstrated a better approach to the pathology, as well as better results in terms of both vital prognosis, but also in terms of quality of life (disability, logical disorders, etc.). However, this treatment modality remains little known to the general public, and generates a high level of anxiety for patients.
  The anxiety of these patients could be reduced by the addition of a paramedical consultation and the use of a flow model to explain and visualize the procedure.
  The study will include 72 patients per group (i.e. a total of 144 patients, with a 10% loss of blood pressure) to achieve a two-point reduction in the anxiety score measured by the APAIS grid.
  Arms: Experimental

SUMMARY:
Intracranial aneurysm is a malformation of the cerebral arteries, identifying with a focal dilatation of the wall of an intracranial artery. This pathology is a fragility of the arterial wall which dilates abnormally creating ≪ a pocket ≫ where blood circulates under pressure. Due to their parietal fragility, aneurysms can grow or rupture. In addition, certain factors such as chronic arterial hypertension, smoking and chronic alcohol intoxication favor the risk of aneurysm rupture or growth. Cerebral aneurysm rupture has a serious prognosis: 10% of patients die before reaching hospital, 25% die within 24 hours, and 40-49% die within 3 months. Interventional neuroradiology offers treatment via an endovascular approach, by obstructing the aneurysm with coils and stents navigating within the arteries. This operation is not without risk of death or per-procedural stroke. In France, it is estimated that 5 to 7 patients per 100,000 of the population suffer a ruptured aneurysm, which means around 5,000 new cases every year. This figure does not take into account patients who die before accessing medical services.

Interventional neuroradiology is a little-known discipline. Lack of knowledge about the activity, the professionals involved and the technologies involved, leads to anxiety among patients.

Moreover, neurological pathologies are often physically undetectable. The investigators note a high degree of anxiety among patients on arrival at the department.However, it is difficult to explain the examination without support.That's why it would be interesting to build a simulation tool.

The investigators note a high degree of anxiety among patients on arrival at the department. However, it is difficult to explain the examination without support. That's why it would be interesting to build a simulation tool.

simulation tool to help explain the procedure: a 3D printer model of the vessels of a full-scale silicone model called the flow model, to be presented at the paramedical consultation for the experimental group. This will enable the patient to visualize the procedure and play an active role in it. The patient will therefore be able to benefit from all the information the procedure and the practices involved, understanding not only how the puncture is made and where, but also how it is arrived at. the aneurysm and how it is treated. In addition, visualizing the procedure will help patients to avoid the unknown, and make it easier to manage their anxiety.

The flow model enables visualization of aneurysmal pathology in a simplified, concrete and didactic way for patients and the general public.

At present, flow models of cerebral aneurysms have already been evaluated by some teams with a view to improving the information provided to the patient, in a non-randomized fashion and partially covering the operation.

To our knowledge, there is no flow model reproducing the entire endovascular operative pathway from the puncture site (femoral or radial approach), the aorta and the graft to the aorta.

the aorta, then the cervical arteries through to the cerebral aneurysm, has yet to be created and used.

The major advantage of this modelization would be to simulate the entire procedure during the consultation, from puncture to placement of the stent and coils occluding the aneurysm. This project is particularly innovative, as it enables the patient to rationalize the procedure, potentially reducing his or her state of anxiety, and putting the patient and paramedical team in a practical situation to face up to the inherent risks of the operation. In addition, flow model simulation will enable the paramedical team to be trained in the practice of interventions. The ANXIFLOW project will therefore form the basis of a new handling training course for the continuing education of radiology technicians.

This will involve preparing the radiology technicians to assist the doctor, preparing the equipment, disinfecting and laying the operating drapes, and anticipating the doctor's needs: prepared coils, micro-catheters, perfusion bag and purge circuit, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patient (aged 18-70) with cerebral aneurysm pathology
* Affiliated to the French social security system
* Patient informed of the study and having signed the informed consent form
* Patient who speaks and understands French

Exclusion Criteria:

* Patient > 70 years of age (benefit/risk balance of preventive treatment against treatment) treatment)
* Patient under guardianship, curatorship, safeguard of justice or legal protection
* Mentally handicapped patient
* Patient with severe psychiatric pathology
* Patient unable to communicate in French
* Patients receiving premedication
* Patient under 18 years
* Blind patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-05-02 (Estimated); Primary Completion 2028-05-02 (Estimated); Study Completion 2028-05-02 (Estimated)

PRIMARY OUTCOMES:
APAIS scale | Before and after paramedical consultation (Day less 7)
  To compare the level of preoperative anxiety according to the APAIS scale before and after the preoperative paramedical consultation between a group of patients receiving standard information (control group) and a group of patients who also benefited from the flow model surgical simulation (experimental group).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah HEMERY, Principal Investigator — CHU CAEN
Locations (1):
- CHU Caen, Caen, France, France